CLINICAL TRIAL: NCT00180947
Title: Phase II Study of Vinorelbine + Cyclofosfamide Association Among Patients Reached of Refractory Tumours or in Relapse
Brief Title: Study of Vinorelbine and Cyclofosfamide Among Patients With Refractory Tumours or in Relapse
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAVE-CYCLO
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Rhabdomyosarcomas; Neoplasms, Connective and Soft Tissue; Ewing Tumor; Osteosarcomas; Neuroblastomas; Medulloblastomas
Keywords: Soft parts tissue
MeSH Terms: conditions — Rhabdomyosarcoma; Neoplasms, Connective and Soft Tissue; Sarcoma, Ewing; Osteosarcoma; Neuroblastoma; Medulloblastoma | interventions — Vinorelbine

INTERVENTIONS:
Drug: Vinorelbine, cyclofosfamide

SUMMARY:
This is a phase II study to determine the antitumor activity of Vinorelbine and Cyclofosfamide association among patients with refractory tumours or in relapse with rhabdomyosarcomas and other soft tissue tumours, Ewing tumours, osteosarcomas, neuroblastomas or medulloblastomas.

ELIGIBILITY:
Inclusion Criteria:

* Age > 12 months and < 25 years
* Measurable disease
* Score of Lansky > 30 or World Health Organization (WHO) score < 2
* Life expectancy > 2 months
* Satisfactory hematologic conditions:

  * Polynuclear neutrophiles > 1 X 10^9/l.
  * Platelets > 100 X 10^9/l or > 50 X 10^9 in the event of medullary invasion.
* Creatinine < 1.5 of normal for age or clearance > 70 ml/min/1.73 m2
* Normal hepatic function:

  * Bilirubin < 3 N
  * ASAT and ALAT < 2,5 N).
* Absence of toxicity of bodies (Rank > 2 according to coding National Cancer Institute-Common Toxicity Criteria [NCI-CTC] version 2.0)
* Absence of antecedent of hematuric cystitis to repetition
* Written consent, signed by the patient or the two parents or holder(s) of the parental authority of the minor subjects

Exclusion Criteria:

* Does not satisfy the criteria of eligibility

Ages: 12 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210
Dates: Start 2003-06

PRIMARY OUTCOMES:
To determine the antitumor activity of Vinorelbine and oral Cyclofosfamide association in refractory tumours or in relapse

SECONDARY OUTCOMES:
To evaluate the hematologic tolerance of this association
To evaluate the pharmacokinetics of injectable Vinorelbine

CONTACTS AND LOCATIONS:
Overall Officials: Odile OBERLIN, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave-Roussy, Villejuif, France